CLINICAL TRIAL: NCT02600975
Title: A Phase I Study to Assess the Safety and Immunogenicity of a Protein Particle Malaria Vaccine Candidate, R21, Administered With AS01B in Healthy UK Volunteers
Brief Title: A Study to Assess the Safety and Immunogenicity of a Malaria Vaccine Candidate, R21, Administered With AS01B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC056
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): 10µg of R21 with AS01B on days 0, 28, and 56.
  Interventions: Biological: R21 with ASO1B
- Group 2 (Active Comparator): 50µg of R21 with AS01B on days 0, 28, and 56.
  Interventions: Biological: R21 with ASO1B

INTERVENTIONS:
Biological: R21 with ASO1B — R21 with ASO1B

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered an experimental malaria vaccine, R21. The R21 vaccine will be administered with the adjuvant AS01B.

All vaccinations will be administered intramuscularly. Each volunteer will receive three vaccinations in total.

There are two different vaccine schedules:

Group 1 will receive R21 10µg with AS01B on days 0, 28, and 56. Group 2 will receive R21 50µg with AS01B on days 0, 28, and 56.

The study will assess the safety of the vaccine, and the immune responses to the vaccination. Immune responses are measured by tests on blood samples.

Healthy adult volunteers will be recruited in Oxford and Southampton, England.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational malaria vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* History of clinical malaria (any species)
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of administration of R21 with adjuvant AS01B. This will be done by recording the number of participants who experience adverse events, and the severity of any adverse events. | 34 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - CCVTM, University of Oxford, Oxford
  - NIHR Wellcome Trust Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: Undecided
Yes when manuscript is published